CLINICAL TRIAL: NCT05954052
Title: An Open-Label Study of Glutathione in Children With Autism Spectrum Disorder
Brief Title: A Study of Glutathione in Children With Autism Spectrum Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding and difficulty with phlebotomy in children with Autism
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB19-0017
Record Dates: First submitted 2023-05-18; First posted 2023-07-20 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Glutathione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Glutathione Oral Supplementation (Experimental): Glutathione will be the only study medication dispensed to subjects for this study. Subjects will be told to take the first dose of study medication after breakfast each day and the second dose in the evening after dinner. The proposed dose range for Glutathione in this study will be 1000mg-3000mg/day based on the subject's weight.
  Interventions: Drug: Glutathione

INTERVENTIONS:
Drug: Glutathione — Giving supplement orally

SUMMARY:
The aim of this study is to investigate if taking a supplement called Glutathione by mouth is safe and practical for children and teenagers with Autism Spectrum Disorder (ASD). The researchers plan to involve 24 individuals with ASD and give them oral Glutathione for 12 weeks.

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the safety and feasibility of oral Glutathione in children and adolescents who have Autism Spectrum Disorder. Twenty-four subjects with ASD will receive 12 weeks of oral Glutathione reduced. The hypothesis to be tested is that: Oral Glutathione will be effective in increasing the blood level of Glutathione, which may help to decrease some problem behaviors and irritability in this particular ASD population. The second aim of this study is to evaluate the tolerability of oral Glutathione. The proposed study may provide needed data for future studies aimed at the treatment of aggressive behaviors that can be seen in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ages 4-17
* Current diagnosis of Autism Spectrum Disorder as determined by criteria in DSM-5
* Parents of Children ages 4-17 with a current diagnosis of Autism Spectrum Disorder as determined by criteria in DSM-5

Exclusion Criteria:

* Unstable medical illness or clinically significant abnormalities on physical examination;
* History of seizures;
* History of Hematological disorders;
* Myocardial infarction within 6 months;
* Current pregnancy or lactation, or inadequate contraception in girls of childbearing potential;
* Current or recent (past 3 months) DSM-5 substance abuse or dependence;
* Illegal substance use within 2 weeks of study initiation;
* Previous treatment with Glutathione;
* Current treatment with N-acetylcysteine, milk thistle, Vitamin C, Vitamin B, Grape Seed Extract, Amino Acids, or Zinc
* Current treatment with Dextromethorphan, D-cycloserine, Amantadine, Memantine, Lamotrigine or Riluzole
* Asthma

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karam Radwan, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following the completion of the trial and until 2 years from the publication of the trial outcome data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glutathione Oral Supplementation
Started | 6
Completed | 5
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Glutathione Oral Supplementation
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.67 [10 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Aberrant Child Checklist, Looking at Change in the Subscale of the ABC
Description: The Aberrant Behavior Checklist (ABC) measures psychiatric symptoms and behavioral disturbances in individuals with IDD across five subscales: Irritability (0-45), Social Withdrawal (0-48), Stereotypic Behavior (0-21), Hyperactivity (0-48), and Inappropriate Speech (0-12). Each subscale score is summed to calculate a total score ranging from 0 to 174. Higher scores indicate worse outcomes, with no specific cutoff values, as the measure is used alongside diagnostic tools like the Autism Diagnostic Observation Schedule (ADOS). The ABC is designed to establish baseline symptoms and monitor changes over time, where a decrease in scores reflects improvement, and an increase indicates worsening symptoms.The Aberrant Behavior Checklist (ABC) consists of five subscales: Irritability (0-45), Lethargy (0-48), Stereotypic Behavior (0-21), Hyperactivity (0-48), and Inappropriate Speech (0-12). Higher scores represent more severe symptoms. The total ABC score ranges from 0 to 174
Time Frame: baseline and 12 weeks. To clarify, all pre-specified Primary and Secondary Outcome Measures were collected at baseline and the 12-week endpoint only. No intermediate assessments were conducted.
Population: All participants who received at least one dose of oral glutathione and had both baseline and Week 12 (or endpoint) Aberrant Behavior Checklist (ABC) assessments available (n=5). One participant discontinued after 2 weeks due to increased irritability and was excluded from the change analysis
Measure: Mean (62% Confidence Interval); unit: units on a scale
Groups:
- Glutathione: We have one arm who took supplement
Arm/Group | Glutathione
Number analyzed (Participants) | 5
units on a scale
  ABC: Irritability | 18.60 [15.56 to 20.64]
  ABC: Lethargy | 14.40 [10.99 to 17.81]
  ABC: Stereotypy | 8.80 [7.01 to 10.59]
  ABC: Hyperactivity | 14.80 [13.25 to 16.35]
  ABC: Inappropriate Speech | 6.40 [5.12 to 7.68]
Statistical Analysis 1: Comparison: Glutathione; For the analysis of (ABC) scores at baseline and 12 weeks in this single-arm, open-label pilot study (n=6 participants, all with paired data including the early dropout), we use superiority test, This aligns with the study's hypothesis that oral glutathione supplementation would lead to an improvement (i.e., a decrease in ABC scores, indicating reduced irritability). Superiority testing evaluates whether the post-treatment mean (or median) is significantly lower than the baseline; Test type: Superiority; p = 0.1807, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 4, 95% CI 2-sided [-6.24 to 14.24], Standard Deviation 9

2. Secondary Outcome: Social Responsiveness Scale
Description: The Social Responsiveness Scale, Second Edition (SRS-2) is a 65-item caregiver-rated questionnaire that measures the severity of social impairments associated with autism spectrum disorder (ASD) in children and adolescents (ages 2 years 6 months to 18 years). It assesses five domains: Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests and Repetitive Behavior, as well as a Total Score.
  T-scores typically range from approximately 30 to 90+, with scores capped at 90 in cases of severe impairment.
  Higher T-scores indicate greater severity of social impairment (worse outcome), while lower T-scores indicate fewer social difficulties (better outcome).
  Clinically Relevant Thresholds
  T-score ≤ 59: Within normal limits T-score 60-65: Mild range (borderline, subclinical difficulties) T-score 66-75: Moderate range (clinically significant impairment) T-score ≥ 76: Severe range (marked impairment)
Time Frame: We only have the Social Responsiveness Scale measurement at baseline.
Population: All participants who were enrolled and completed the baseline Social Responsiveness Scale (SRS) assessment (n=6)
Measure: Median (Inter-Quartile Range); unit: T-score for this instrument.
Arm/Group | Glutathione Oral Supplementation
Number analyzed (Participants) | 6
T-score for this instrument.
  Social Awareness | 75.5 [58.25 to 86.75]
  Social Cognition | 85.0 [78.5 to 89.25]
  Social Communication | 90.00 [64.5 to 90]
  Social Motivation | 82.0 [75.0 to 83.75]
  Autism Mannerisms | 89.0 [77.5 to 89.75]
  Total Severity | 89 [73.0 to 90]

3. Other Pre Specified Outcome: Change in Clinical Global Impression Scale
Description: The Clinical Global Impression (CGI) is a clinician-rated instrument developed for use in NIMH-sponsored clinical trials to provide a brief global assessment of illness severity, improvement, and therapeutic efficacy. The three commonly reported CGI scales are:
  CGI-Severity (CGI-S): Rates current illness severity from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients).
  CGI-Improvement (CGI-I): Rates change in clinical status from baseline on a 7-point scale, ranging from 1 (Very much improved) to 7 (Very much worse).
  CGI-Efficacy Index (CGI-E): Balances therapeutic efficacy with adverse effects, rated on a 4 × 4 grid, where higher scores reflect minimal efficacy and/or significant side effects.
  Lower CGI-S and CGI-I scores indicate better outcomes (less illness severity and/or greater improvement).
  Higher CGI-E scores reflect worse outcomes (limited efficacy and/or significant side effects).
  Higher CGI-E scores reflect worse outcomes
Time Frame: At baseline and the end of the trial (12 weeks)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Glutathione Oral Supplementation
Number analyzed (Participants) | 6
score on a scale
  Pre-Treatment CGI Severity | 4 [3.25 to 4.75]
  Post-Treatment CGI Severity | 4.5 [3.25 to 5]
  CGI Improvement | 3 [3 to 3.75]
  Efficacy Index | 9 [9 to 11.25]

4. Post Hoc Outcome: Clinical Global Impression - Severity Scale (CGI-S) Range for Participants
Description: Pre-treatment CGI-S ratings ranged from 2 (borderline ill) to 5 (markedly ill). One subject's CGI-S changed from 4 (moderately ill) to 5 (markedly ill); others had no change.
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Post Hoc Outcome: Clinical Global Impression - Improvement Scale: Rates Change in Clinical Status From Baseline on a 7-point Scale, Ranging From 1 (Very Much Improved) to 7 (Very Much Worse).
Description: 1 subject scored 4 (no change), four scored 3 (minimally improved), and one scored 6 (much worse).
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Post Hoc Outcome: CGI-Efficacy Index (CGI-E): Balances Therapeutic Efficacy With Adverse Effects, Rated on a 4 × 4 Grid, Where Higher Scores Reflect Minimal Efficacy and/or Significant Side Effects.
Description: two patients had no therapeutic changes, four had minimal efficacy, five had no side effects, and one dropped out due to significant side effects
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: collected using interview with the family and patient
Arm/Group | Glutathione
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glutathione (N=6)
1 (Nervous system disorders) | 1 (1) — one subject had increased irritability and agitation which was resolved after D/C the supplement
irritability (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glutathione (N=6)
1 (Nervous system disorders) | 1 (1) — increase irratbility

LIMITATIONS AND CAVEATS:
Early termination due to lack of funding and difficulty with phlebotomy in children with Autism

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT05954052/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT05954052/ICF_001.pdf